CLINICAL TRIAL: NCT02475200
Title: Phoenix Post-Approval Registry - Using the Phoenix Atherectomy Systems
Status: Completed | Type: Observational
Sponsor: Volcano Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 150201
Record Dates: First submitted 2015-04-08; First posted 2015-06-18 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Peripheral Arterial Disease; Claudication; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Chronic Limb-Threatening Ischemia | interventions — Atherectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Atherectomy — Selectively cut and remove atheromatous plaque in the lower extremities. Debulking and removal of atherosclerotic burden plaque with Phoenix Atherectomy System.

SUMMARY:
The Phoenix Post-Approval Registry is a prospective, multi-center, single arm registry sponsored by Volcano Corporation to evaluate the short and long term performance and clinical outcomes of the Phoenix Atherectomy System.

DETAILED DESCRIPTION:
The Phoenix Post-Approval Registry is an prospective, multi-center, single arm registry, sponsored by Volcano Corporation, to evaluate the short and long term performance and clinical outcomes of the Phoenix Atherectomy System. The study includes consecutive patients treated with the Phoenix Atherectomy System in a post-market (commercial device use) setting. Patients will be followed under real-world conditions for up to 12 months after the index procedure.

All patients with a planned endovascular revascularization procedure receiving treatment with the Phoenix Atherectomy System as all or part of their PAD treatment strategy may be included. Written informed consent must be obtained from each patient prior to enrollment in the study. Enrolled patients will undergo PAD treatment that includes Phoenix atherectomy, according to institutional or local standard of care. Data collection will include medical record review of procedures performed according to standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is ≥18 years of age.
2. Patient understands the research nature of the study and is willing and capable of providing written informed consent.
3. Scheduled for and receives treatment with the Phoenix Atherectomy System as all or part of their PAD treatment.
4. Meets Phoenix Atherectomy System catheter Instruction for Use (IFU) criteria.

Exclusion Criteria:

* Patients who have ANY of the following exclusion criteria are NOT eligible for the study:

  1. Patients unwilling or unable to comply with the protocol including 12-month follow-up for patients with CLI at baseline.
  2. Patient is participating in another device or drug clinical trial that interferes with this protocol follow up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients who are scheduled to receive atherectomy with the Phoenix Atherectomy System used according to local standards.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2018-04-08 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Phoenix device performance | 30 days
  Rates of TECHNICAL SUCCESS (ratio of Phoenix treated lesions with <=50% residual diameter stenosis to all Phoenix treated lesions); and PROCEDURAL SUCCESS (ratio of target lesion residual stenosis of <=30% after treatment with Phoenix and adjunctive treatments to all treated lesions)

SECONDARY OUTCOMES:
Ankle brachial index (ABI) | 12 months
  Change in ABI between baseline and 12-month follow-up visits in patients with CLI at baseline
Society for Vascular Surgery's Wound, Ischemia, and foot Infection (WIfI) category | 12 months
  Change in WIfI category between baseline and 12-month follow-up visits in patients with CLI at baseline
Rutherford Clinical Category | 12 months
  Change in Rutherford Clinical Category between baseline and 12-month follow-up visits in patients with CLI at baseline
Clinically-driven target vessel revascularization (TVR) in patients with CLI at baseline | 12 months
  Rate of repeat percutaneous (endovascular) or surgical intervention to treat objectively documented signs/symptoms of recurrent ischemia attributable to the target vessel at a site other than the index lesion(s)
Clinically-driven target lesion revascularization (TLR) in patients with CLI at baseline | 12 months
  Rate of repeat percutaneous (endovascular) or surgical intervention to treat objectively documented signs/symptoms of recurrent ischemia attributable to the index lesion(s)
Unplanned target limb amputation in patients with CLI at baseline | 30 days
  Rate of amputation associated with the target limb that occurs between the index procedure and 30 days that was not previously planned as part of the overall treatment strategy
Unplanned target limb amputation in patients with CLI at baseline | 12 months
  Rate of amputation associated with the target limb that occurs between the index procedure and 12 months that was not previously planned as part of the overall treatment strategy

CONTACTS AND LOCATIONS:
Overall Officials: Bradley S Matsubara, MD, Study Director — Volcano Corporation
Locations (5):
- United States (5):
  - Pima Vascular, Tucson, Arizona
  - St. John Hospital, Detroit, Michigan
  - Mid-Michigan Heart & Vascular Center, Saginaw, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - Cardiovascular Specialists of Texas, Austin, Texas